CLINICAL TRIAL: NCT06633224
Title: An Evaluation of Changes in the Relationships Between Fatigue and Molecular Mechanisms in Cancer Patients Receiving Curative-Intent Combined Chemotherapy and Radiation Therapy (CCRT)
Brief Title: Fatigue and Molecular Mechanisms in Cancer Patients Receiving CCRT
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 239814; R37CA233774 (NIH); NCI-2024-08455 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Thoracic Cancer; Gynecologic Cancer; Head and Neck Cancer; Gastrointestinal Cancer
Keywords: Basic Science Research
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms | interventions — Blood Specimen Collection; Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 16 mL of blood and a stool sample will be obtained at each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer Patients: Participants will have blood and stool samples collected within 5 days of any pre or post treatment timepoint prior to, during, at completion of therapy and up to 34 weeks following non-investigational, standard of care, CCRT. Participants will also be given quality of life questionnaires to complete throughout the course of the study.
  Interventions: Procedure: Blood Specimen Collection; Other: Stool Specimen Collection; Other: Quality of Life (QOL) Questionnaires

INTERVENTIONS:
Procedure: Blood Specimen Collection — Blood samples will be obtained throughout the course of the study
  Other Names: Blood Specimen
Other: Stool Specimen Collection — Stool samples will be obtained throughout the course of the study
  Other Names: Stool Specimen
Other: Quality of Life (QOL) Questionnaires — Surveys will be given throughout the course of the study.
  Other Names: Quality of Life Surveys

SUMMARY:
Cancer-related fatigue (CRF) is a significant problem for cancer patients. This prospective, basic science, observational study will evaluate for changes in CRF associated with molecular characteristics prior to, during, and at the completion of non-investigational, standard-of-care, combined chemotherapy and radiation therapy (CCRT) and to develop and assess predictive models for CRF severity.

DETAILED DESCRIPTION:
Primary Objective For mean, morning and evening CRF:

Aim 1. Evaluate for associations between phenotypic characteristics and initial levels and the trajectories of CRF.

Aim 2. Evaluate for associations between changes in CRF severity and changes in gene expression levels prior to the initiation and at the end of CCRT.

Aim 3. Evaluate for associations between changes in CRF severity and changes in circulating free cytokine levels prior to the initiation and at the end of CCRT.

Aim 4. Develop and assess predictive models for CRF severity midway, at the end of, and at least six months post-CCRT using demographic, clinical, and molecular characteristics collected prior the initiation of CCRT.

Secondary Objectives For the commonly co-occurring symptom of chemotherapy-induced peripheral neuropathy (CIPN):

Secondary Aim 5. Evaluate for associations between phenotypic characteristics and initial levels and the trajectories of CIPN.

Secondary Aim 6. Evaluate for associations between changes in CIPN severity and changes in gene expression levels prior to the initiation and at the end of CCRT.

Secondary Aim 7. Evaluate for associations between changes in CIPN severity and changes in circulating free cytokine levels prior to the initiation and at the end of CCRT.

Secondary Aim 8. Develop and assess predictive models for CIPN severity midway, at the end of, and at least six months post-CCRT using demographic, clinical, and molecular characteristics collected prior the initiation of CCRT.

Exploratory Aim 1 - Evaluate the feasibility of the protocol for the collection of stool samples.

Exploratory Aim 2 - Evaluate the feasibility of processing and storing stool samples.

Exploratory Aim 3 - Evaluate the feasibility of processing and storing performing blood samples and performing Cytometry by time of flight (CyTOF) assays.

ELIGIBILITY:
Inclusion Criteria:

* Participants have not received any prior treatment (i.e., cancer systemic therapies or radiation therapy) in the month except surgery or inductive Chemotherapy (CTX).
* Participants receiving >= 15 fractions.
* Participants is male or female and is >18 years of age on the day of signing the informed consent.
* Ability to understand a written informed consent document.
* Able and willing to complete all of the study questionnaires and provide blood and stool samples prior to, midway, and following the completion of treatment.
* Willing to have medical records reviewed for clinical information.
* Able to read, write and understand English or Spanish.

Exclusion Criteria:

* Contraindication to phlebotomy for removal of approximately 50 mL of peripheral blood within 6 week period (Institutional Review Board (IRB) limit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients willing to travel to San Francisco, receiving CCRT at University of California, San Francisco (UCSF) for cancers of the head and neck, gynecological, gastrointestinal, or thoracic sites.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Measure associations between changes in cancer-related fatigue (CRF) and changes in gene expression over time | Up to 34 weeks
  Association between phenotypic characteristics and initial levels and trajectories of CRF severity will be assessed using a hierarchical linear model (HLM) approach.
Measure associations between changes in CRF and changes in cytokine levels over time | Up to 34 weeks
  Association between changes in CRF severity and biomarker levels prior to the initiation and at the end of CCRT. Linear regression will be used to evaluate for associations between fatigue changes and biomarker levels at baseline controlling for covariates identified in the initial primary outcome. Adjustments for multiple comparisons will be conducted using the Benjamini-Hochberg (BH) procedure at a false discovery rate (FDR) of 10%.
Measure associations between changes in CRF and changes in gene expression over time | Up to 34 weeks
  Association between changes in CRF severity and gene expression prior to the initiation and at the end of CCRT. Linear regression will be used to evaluate for associations between fatigue changes and biomarker levels at baseline controlling for covariates identified in the initial primary outcome. Adjustments for multiple comparisons will be conducted using the Benjamini-Hochberg (BH) procedure at a false discovery rate (FDR) of 10%.
Evaluate the predictive utility of gene expression and cytokine data | Up to 34 weeks
  A validated prediction model of CRF severity will be generated using machine learning (ML) methods to minimize the error between predicted and observed levels of fatigue midway through CCRT, at the completion of CCRT, and at least six months following the completion of CCRT. Evaluation of common ML algorithms for prediction accuracy and evaluation of model performance as compared to simple linear regression. Separate training and testing sets will be created, cross-validated, and repeated and impact of each variable will be determined.

SECONDARY OUTCOMES:
Evaluate for associations between changes in chemotherapy-induced peripheral neuropathy (CIPN) and changes in gene expression | Up to 34 weeks
  The association between phenotypic characteristics and initial levels and trajectories of CIPN severity will be evaluated using a hierarchical linear model (HLM) approach.
Evaluate for associations between changes in CIPN and changes in cytokine levels | Up to 34 weeks
  The association between phenotypic characteristics and initial levels and trajectories of CIPN severity will be evaluated using a hierarchical linear model (HLM) approach.
Evaluate the predictive utility of gene expression and severity of CIPN | Up to 34 weeks
  The association between changes in CIPN severity and gene expression prior to the initiation and at the end of CCRT. Linear regression will be used to evaluate for associations between CIPN changes and gene expression at baseline controlling for covariates identified in previous objectives/endpoints. Adjustments for multiple comparisons will be performed using the Benjamini-Hochberg (BH) procedure at a false discovery rate (FDR) of 10%.
Evaluate the predictive utility of cytokine levels and severity of CIPN | Up to 34 weeks
  The association between changes in CIPN severity and cytokine levels prior to the initiation and at the end of CCRT. Linear regression will be used to evaluate for associations between CIPN changes and cytokine levels at baseline controlling for covariates identified in previous objectives/endpoints. Adjustments for multiple comparisons will be performed using the Benjamini-Hochberg (BH) procedure at a false discovery rate (FDR) of 10%.
Evaluate the predictive model of severity of CIPN | Up to 34 weeks
  The predictive utility will be assessed through a validated prediction model of CIPN severity using machine learning (ML) methods to minimize the error between predicted and observed levels of CIPN midway through CCRT, at the completion of CCRT, and at least six months following the completion of CCRT. We will evaluate common ML algorithms for prediction accuracy and evaluate their performance as compared to simple linear regression

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No